CLINICAL TRIAL: NCT05997602
Title: A Multi-center, Open-label, Single Arm Phase 2 Study to Evaluate the Efficacy, Safety, and Pharmacokinetic Characteristics of FCN-159 in Pediatric Patients With Refractory/Recurrent Langerhans Cell Histiocytosis
Brief Title: To Evaluate the Efficacy, Safety, and PK Characteristics of FCN-159 in Pediatric Patients With Refractory/Recurrent LCH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCN-159-004
Record Dates: First submitted 2023-08-08; First posted 2023-08-18 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Langerhans Cell Histiocytosis; LCH
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCN-159 (Experimental): Experimental: FCN-159 Dosage form:tablet Specification: 1mg，4mg Dose: FCN-159 5mg/m² (Maximum dose does not exceed 8mg), orally, once daily
  Interventions: Drug: FCN-159

INTERVENTIONS:
Drug: FCN-159 — 5mg/m² (Maximum dose does not exceed 8mg, the recommended oral dose for adults), orally, once daily, continuously for 28 days per cycle.

SUMMARY:
This is a rare disease, single-arm, open-label,multi-center, non-randomized Phase 2 clinical study to evaluate the efficacy, safety, and pharmacokinetic characteristics of FCN-159 monotherapy in pediatric patients with refractory/recurrent Langerhans cell histiocytosis (LCH).

DETAILED DESCRIPTION:
This is a rare disease, single-arm, open-label,multi-center, non-randomized Phase 2 clinical study to evaluate the efficacy, safety, and pharmacokinetic characteristics of FCN-159 monotherapy in pediatric patients with refractory/recurrent Langerhans cell histiocytosis (LCH). Approximately 56 pediatric patients will be enrolled in this study.The study included screening period, treatment period and follow-up period. Subjects will receive FCN-159 5mg/m² (NMT 8mg, the recommended oral dose for adults), orally, once daily, continuously for 28 days per cycle. Subjects will be treated until disease progression (PD), intolerable toxicity, withdrawal of consent, death, or other protocol-specified reasons. According to the PET Response Criteria and Langerhans Cell Histiocytosis Evaluation and Treatment Guidelines, tumor assessment will be performed until disease progression, death, and withdrawal of information Intention, loss of follow-up, initiation of new antitumor therapy, or study termination.Efficacy evaluation will be performed by the investigator and the Independent Review Committee (IRC), respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-16 (inclusive)
2. Patients with histologically confirmed Langerhans cell histiocytosis (LCH) diagnosed by the central laboratory.
3. If sufficient tumor tissue samples and peripheral blood samples are available, central laboratory biomarker testing is required as follows: including but not limited to ERBB3, BRAF, ARAF, HRAS, KRAS, NRAS, MEK (MAP2K1 and MAP2K2), and other MEK upstream genes.If inability to get tissue, the gene testing results from a local laboratory also can be accepted.
4. Patients who have received at least prior first-line systemic treatment, defined as treatment including vinblastine (VBL) and glucocorticoids for at least 2 weeks. VBL can be substituted with vincristine (VCR) or vindesine (VDS). Alternatively, patients may be unable to tolerate chemotherapy due to severe chemotherapy toxicity. Inability to tolerate chemotherapy is defined as one of the following: Severe liver impairment (liver enzyme elevation ≥ 5 × upper limit of normal (ULN) and bilirubin elevation ≥ 1.5 × ULN), severe neurotoxicity related to vinca alkaloids, chemotherapy-related intracranial hypertension, or grade 4 bone marrow depression with severe infection (sepsis, severe pneumonia, etc.) after chemotherapy.
5. Refractory/relapsed LCH is defined as the presence of one of the following:

   1. Failure of prior treatment, i.e., no regression in risk organs after at least 2 weeks of systemic treatment, or overall evaluation of AD-progression or AD-mix;
   2. Initial response of the disease to first or second-line systemic treatment is NAD or AD-better or AD-stable, followed by disease reactivation after maintenance therapy for more than 3 months. Second-line treatment includes cytarabine and/or cladribine.
   3. Persistent mutated gene positive in plasma free DNA testing during prior treatment (confirmed by 2 consecutive tests) or retest positive after treatment discontinuation;
   4. Lack of regression in the affected central nervous system (including the pituitary gland) after treatment;
   5. Presence of bone marrow involvement and/or hemophagocytic lymphohistiocytosis (HLH);
6. Presence of evaluable lesions based on PET response criteria (PRC).
7. Patients who have to have recovered from all acute toxic effects of prior anti-tumor therapy, and all relevant toxicities must be ≤ grade 1 (except for alopecia and ototoxicity).
8. Expected survival at least ≥ 3 months;
9. Lansky (≤ 15 years old) and Karnofsky (≥ 16 years old) performance status scores should be ≥ 50%, as shown in Appendix 4.
10. Patients or their legal guardians must be able to understand and willingly sign a written informed consent form.
11. For women of childbearing potential, a serum human chorionic gonadotropin (HCG) pregnancy test must be negative within 7 days before starting treatment.
12. For female patients of childbearing potential: Patients should agree to use effective contraception methods during the treatment period and for at least 90 days after the last dose of study treatment, using dual barrier contraception methods such as condoms, oral or injectable contraceptives, intra-uterine contraceptive devices, etc. Male patients should agree to refrain from donating sperm for at least 90 days after the last dose of study treatment.
13. Adequate bone marrow function: Absolute neutrophil count ≥ 1.0×10^9/L, hemoglobin ≥ 90g/L, and platelets ≥ 75×10^9/L without the use of blood transfusions, blood products, or granulocyte colony-stimulating factors. Patients with hematocytopenia below these thresholds due to the underlying disease may be considered for inclusion based on the investigator's comprehensive judgment.
14. Adequate hepatic and renal function: Serum total bilirubin ≤ 1.5 × the upper limit of normal (ULN), or ≤ 5× ULN for patients with Gilbert's syndrome or liver involvement; aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (AKP) ≤ 2.5 × ULN, or ≤ 10 × ULN for patients with liver involvement; albumin ≥ 3g/dL; and creatinine clearance or isotopic glomerular filtration rate (GFR) ≥ 50ml/min/1.73㎡or serum creatinine based on age; hepatic and renal impairment caused by the primary disease may be considered for inclusion based on the investigator's comprehensive judgment.
15. Coagulation: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN.

Exclusion Criteria:

1. Patients who have received any of the following prior treatments:

   1. Chemotherapy, targeted therapy, immunotherapy, biologic therapy, or herbal anti-tumor therapy for LCH within 4 weeks or < 5 half-lives (whichever is shorter)before the start of the study drug .
   2. Strong CYP3A4, CYP2C8, and CYP2C9 inhibitors or inducers within 14 days before the start of the study drug, except for topical skin application.
   3. Gowth factors that promote platelet or white blood cell count or function within 7 days before the start of the study drug.
   4. Radiotherapy or major surgical treatment (including craniotomy, thoracotomy, laparotomy, open bone or joint surgery, etc.) within 4 weeks before the start of the study drug.
   5. Participated in other interventional clinical trials within 4 weeks before the start of the study drug.
   6. MEK 1/2 inhibitors (those who have received this treatment for a short period of ≤ 2 weeks may be included).
   7. Anticoagulants within 7 days before the start of the study drug for patients with brain tumors (intracranial masses).
   8. Prednisone treatment < 0.5mg/kg/day (or equivalent dose of other corticosteroids) is allowed within one month before enrollment, but must be discontinued 14 days before the start of the study drug. Patients with brain lesions receiving corticosteroid therapy for brain edema must maintain a stable dose for 14 days before enrollment. Hormone replacement therapy is allowed for patients with hypopituitarism due to primary disease involvement of the pituitary.
2. Patients with a history of other malignant tumors or concurrent other malignant tumors (excluding cured non-melanoma skin basal cell carcinoma, ductal carcinoma in situ of the breast, or cervical carcinoma in situ).
3. Uncontrolled hypertension (with medication treatment): Blood pressure (BP) greater than or equal to the 95th percentile for age, height, and sex, as described in Appendix 6.
4. Patients with dysphagia, active gastrointestinal disease, malabsorption syndrome, or other conditions that may affect the absorption of the study drug.
5. Prior or current history of retinal vein obstruction (RVO), retinal pigment epithelial detachment (RPED), glaucoma, and other clinically significant abnormal ophthalmologic examination results.
6. Interstitial pneumonia, including clinically significant radiation pneumonitis. Except for interstitial pneumonia caused by pulmonary involvement of the primary disease.
7. Patients will be excluded if their cardiac function or comorbidities meet any of the following criteria:

   1. During the screening period, 12-lead electrocardiogram (ECG) measurements will be taken three times at the study center with a mean value calculated using the QTcF formula provided by the instrument; patients with a mean value of QTcF > 470 milliseconds or with risk factors for QTcF prolongation, such as uncorrected hypokalemia, congenital long QT syndrome, or receiving drugs known to prolong QTcF interval (mainly class Ia, Ic, and III antiarrhythmic drugs) will be excluded from the study. Drugs with the potential to prolong the QTcF interval are listed in Appendix 7.
   2. New York Heart Association (NYHA) Class 2 and above congestive heart failure as shown in Appendix 5.
   3. Clinically significant arrhythmias, including but not limited to complete left bundle branch block, and second-degree atrioventricular block.
   4. Known presence of clinically significant coronary heart disease, cardiomyopathy, or severe valvular disease.
   5. Echocardiography examination indicating left ventricular ejection fraction (LVEF) < 50%.
8. Patients with active bacterial, fungal, or viral infections, including active hepatitis B (defined as positive hepatitis B surface antigen and hepatitis B virus DNA > 1000IU/ml or meeting the diagnostic criteria for active hepatitis B infection at the study center) or hepatitis C (positive hepatitis C virus RNA), or human immunodeficiency virus (HIV positive) infection.
9. Patients with known allergies to the study drug, other MEK1/2 inhibitors, or their excipients.
10. Patients with known tumor tissue genetic testing that indicates the presence of MAP2K1 exon 3 deletions (del) or deletion-insertion type (delins/indels) mutations.
11. The investigator considers clinically significant cases that will impede participation in the study or prevent compliance with safety requirements.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-05-14 (Estimated); Study Completion 2027-05-14 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Evaluated by Independent Review Committee (IRC) Based on PET Response Criteria (PRC) | up to 24months
  ORR Evaluated by Independent Review Committee (IRC) Based on PET Response Criteria (PRC) is defined as the percentage of participants who achieved a best overall response of CMR or PMR assessed by IRC .

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Evaluated by Investigator Based on PET Response Criteria (PRC) and Langerhans Cell Histiocytosis Evaluation and Treatment Guidelines (Histiocyte Society, April 2009, hereinafter referred to as "Guidelines") | up to 24months
  The ORR Evaluated by Investigator Based on PRC is defined as the percentage of participants who achieved a best overall response of CMR or PMR assessed by investigator.
  The ORR Evaluated by Investigator Based on "Guidelines" is defined as the percentage of participants who achieved confirmed NAD or AD-better assessed by investigator.
Disease Control Rate (DCR) Evaluated by Investigator Based on PET Response Criteria (PRC) and "Guidelines". | up to 24months
  The DCR Evaluated by Investigator based on PRC is defined as the percentage of participants who achieved a best overall response of CMR or PMR or SMD assessed by investigator.
  The DCR Evaluated by Investigator Based on "Guidelines" is defined as the percentage of participants who achieved a confirmed NAD or AD-better or AD-stable assessed by investigator.
Clinical benefit rate (CBR) Evaluated by Investigator Based on PRC and "Guidelines". | up to 24months
  The CBR Evaluated by Investigator based on PRC is defined as the percentage of participants who achieved a best overall response of CMR or PMR or SMD for a duration of ≥ 24 weeks assessed by investigator.
  The CBR Evaluated by Investigator Based on "Guidelines" is defined as the percentage of participants who achieved confirmed NAD or AD-better or AD stable for a duration of ≥ 24 weeks assessed by investigator.
Time to Response (TTR) Evaluated by Investigator Based on PET Response Criteria (PRC) and "Guidelines" | up to 24months
  The TTR Evaluated by Investigator based on PRC is defined as the time from the first documented achievement of CMR or PMR (whichever comes first) assessed by investigator.
  The TTR Evaluated by Investigator based on the "Guidelines" criteria is defined as the time from the first documented achievement of NAD or AD-better (whichever comes first) assessed by investigator.
One-year Progressive Free Survival (PFS) Rate Evaluated by Investigator Based on PET Response Criteria (PRC) and "Guidelines" | up to 12months
  The 1-year PFS Rate Evaluated by Investigator based on PRC is defined as the percentage of participants who did not achieve the first documented occurrence of PMD or death (whichever comes first) within one year after first administration of the study drug assessed by investigator.
  The 1-year PFS Rate Evaluated by Investigator based on "Guidelines" is defined as the percentage of participants who did not achieve the first documented occurrence of AD-progression or death (whichever comes first) within one year after first administration of the study drug assessed by investigator.
Progressive Free Survival (PFS) Evaluated by Investigator Based on PET Response Criteria (PRC) and "Guidelines" | up to 24months
  The PFS Evaluated by Investigator based on PRC is defined as the time from the first administration of the study drug to the first documented occurrence of PMD or death (whichever comes first) assessed by investigator.
  The PFS Evaluated by Investigator based on "Guidelines" is defined as the time from the first administration of the study drug to the first documented occurrence of AD-progression or death (whichever comes first) assessed by investigator.
Overall Survival (OS) | up to 24months
  The OS is defined as the time from the first administration of the study drug in patients to death from any cause. Data from the patient without events will be censored at the date the patient is last known to be alive
One-year Overall Survival (OS) Rate | up to 12months
  The 1year OS Rate is defined as as the percentage of participants who did not achieve death due to any cause within one year after first administration of the study drug.
Two-year Progressive Free Survival (PFS) rate Evaluated by the PRC and "Guidelines" | up to 24months
  The 2-year PFS Rate Evaluated by Investigator based on PRC is defined as the percentage of participants who did not achieve the first documented occurrence of PMD or death (whichever comes first) within two year after first administration of the study drug.
  The 2-year PFS Rate Evaluated by Investigator based on "Guidelines" is defined as the percentage of participants who did not achieve the first documented occurrence of AD-progression or death (whichever comes first) within two year after first administration of the study drug.
Two-year Overall Survival (OS) Rate | up to 24months
  The 2 year OS Rate is defined as the percentage of participants who did not achieve death due to any cause within two year after first administration of the study drug.
Treatment-emergent adverse events (TEAEs) | up to 24months
  Type and frequency of treatment-emergent adverse events (TEAEs) with toxicity grades evaluated according to the National Cancer Institute-Common Toxicity Criteria Adverse Event (NCI-CTCAE) version 5.0.
Plasma Concentration of FCN-159 | up to 24months
  Evaluation of the pharmacokinetic characteristics of FCN-159

CONTACTS AND LOCATIONS:
Overall Officials: Rui Zhang, MD, Principal Investigator — Beijing Children's Hospital,Captial Medical University
Locations (11):
- China (11):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Children's Hospital Affiliated to the Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-Sen Memorial Hpsipital,Sun Yat-Sen Unniversity, Guangzhou, Guangdong
  - The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Henan Children's Hospital Zhengzhou Children's Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - West China Second University Hospital,Sihuan University/West China women's and Children's Hospital, Chengdu, Sichuan
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Children's Hospital of Soochow University, Suzhou

IPD SHARING:
Plan to Share IPD: No